CLINICAL TRIAL: NCT06658197
Title: Efficacy and Safety of Tenecteplase Bridging Mechanical Thrombectomy for Acute Large Vessel Occlusive Stroke(TNK-LVO) :a Phase 3, Multicentre, Open-label, Randomised Controlled Trial
Brief Title: Efficacy and Safety of Tenecteplase Bridging Mechanical Thrombectomy for Acute Large Vessel Occlusion Stroke
Acronym: TNK-LVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2024]288-001
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Stroke, Ischemic; Stroke, Acute; Thrombosis, Brain; Drug Effect
Keywords: Ischemic stroke; Tenecteplase
MeSH Terms: conditions — Ischemic Stroke; Stroke; Intracranial Thrombosis | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tenecteplase (Experimental): Subjects assigned to this arm will receive an intravenous bolus of 0.25mg/kg tenecteplase before the mechanical thrombectomy.
  Interventions: Drug: Tenecteplase
- alteplase (Active Comparator): Subjects assigned to this arm will receive an intravenous 0.9 mg/kg alteplase(10% bolus +90% infusion/1 hour) before the mechanical thrombectomy.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase 0.25mg/kg administered as a single rapid intravenous bolus (maximum dose 25mg) plus mechanical thrombectomy
  Other Names: TNK
  Arms: tenecteplase
Drug: Alteplase — Alteplase 0.9 mg/kg administered as 10% bolus +90% infusion/1 hour (maximum dose 90mg) plus mechanical thrombectomy
  Other Names: recombinant tissue plasminogen activator (rtPA)
  Arms: alteplase

SUMMARY:
A phase III, multicentre, prospective, randomised, open-label, blinded-endpoint clinical trial will evaluate two thrombolytic agents for the treatment of acute large vessel occlusion stroke within 4.5 hours from symptoms onset: intravenous tenecteplase bridging mechanical thrombectomy vs. intravenous alteplase bridging mechanical thrombectomy.

DETAILED DESCRIPTION:
Efficacy and Safety of Tenecteplase Bridging Mechanical Thrombectomy for Acute Large Vessel Occlusive Stroke(TNK-LVO) is a phase III, multicenter, prospective, randomized, open-label, blinded-endpoint clinical trial. Randomization will be 1:1 according to reperfusion treatment modalities: (A) Intravenous thrombolysis with tenecteplase (0.25 mg/kg) plus mechanical thrombectomy vs. (B) Intravenous thrombolysis with alteplase (0.9 mg/kg) plus mechanical thrombectomy. For the primary outcome, the subjects will be followed up within 90 days after randomization. The primary outcome will be the Functional independence defined as modified Rankin Score ≤ 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18-80 years.
2. AIS symptom onset ≤4.5 hours, onset time refers to the time the patient was last known to be well. (Recommendation time from thrombolysis to puncture within 60 minutes).
3. Arterial occlusion of the internal carotid artery (ICA), anterior cerebral artery (ACA), posterior cerebral artery (PCA), M1 or M2 segment of the middle cerebral artery (MCA), or basilar artery on computed tomography angiography (CTA) or magnetic resonance angiography (MRA).
4. Prestroke mRS score ≤2.
5. Informed consent from the patient or legally authorised representative.

Exclusion Criteria:

1. Patients diagnosed with hemorrhagic stroke (including intraparenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/extradural hematoma, etc.) or other related conditions identified by CT.
2. Contraindication to imaging examinations involving contrast agent injection.
3. Patients presenting with clinical symptoms of coma (NIHSS Score Item 1a = 3).
4. History of intracranial hemorrhage.
5. History of severe head trauma or stroke within the past 3 months.
6. Intracranial or intraspinal surgery within the past 3 months.
7. Major surgery within the past 2 weeks.
8. Gastrointestinal or urinary tract bleeding within the past 3 weeks.
9. Intracranial tumor, arteriovenous malformation, or giant intracranial aneurysm.
10. Active visceral bleeding.
11. Aortic arch dissection.
12. Arterial puncture at a non-compressible site within the past week.
13. Uncontrolled hypertension despite active antihypertensive treatment: Systolic Blood Pressure > 180 mmHg or Diastolic Blood Pressure > 100 mmHg.
14. Acute hemorrhagic tendency, including platelet count < 100 × 10⁹/L or other conditions.
15. Heparin treatment received within the past 24 hours.
16. For patients on oral anticoagulants: INR > 1.7 or PT > 15 seconds.
17. Use of direct thrombin inhibitors or direct Factor Xa inhibitors within the past 48 hours.
18. Blood glucose < 2.8 mmol/L or > 22.2 mmol/L.
19. Hypodensity affecting > 1/3 of the middle cerebral artery territory or an equivalent proportion of the basilar artery territory on non-contrast CT.
20. Rapidly improving symptoms as determined by the investigator.
21. Participation as a subject in another research study within the past 30 days.
22. Any terminal illness where life expectancy is considered not to exceed 1 year.
23. Any condition where, in the judgment of the investigator, the study treatment might pose a risk to the patient or affect the patient's participation in the study.
24. Pregnant women.
25. Known allergy to the active ingredients (Alteplase, Tenecteplase) or any excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
mRS ≤ 2 at 90 days or no change from baseline | 90 days from baseline
  mRS ≤ 2 at 90 days or no change from baseline

SECONDARY OUTCOMES:
mTICI 2b/3 or absence of retrievable thrombus at initial angiogram | initial angiogram
  mTICI 2b/3 or absence of retrievable thrombus at initial angiogram
mRS at 90 days from baseline | 90 days from baseline
  mRS at 90 days from baseline
mRS 0-1 at 90 days or no change from baseline | 90 days from baseline
  mRS 0-1 at 90 days or no change from baseline
Barthel index at 90 days from baseline | 90 days from baseline
  Barthel index at 90 days from baseline
NIHSS reduce ≥ 8 or reaching 0-1 at 3 days from baseline | 3 days from baseline
  NIHSS reduce ≥ 8 or reaching 0-1 at 3 days from baseline
Change of NIHSS at 1、3、7 days from baseline | 1、3、7 days from baseline
  Change of NIHSS at 1、3、7 days from baseline

OTHER OUTCOMES:
sICH within 36 hours from baseline | 36 hours from baseline
  Defined by Safe Implementation of Thrombolysis in Stroke and The European Cooperative Acute Stroke Study III
Vascular death within 90 days from baseline | Within 90 days from baseline
  Death from stroke, heart attack or pulmonary embolism
Death from any cause within 90 days from baseline | Within 90 days from baseline
  Death from any cause within 90 days from baseline
SAEs within 90 days from baseline | Within 90 days from baseline
  Severe adverse events within 90 days from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhai Guo, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No